CLINICAL TRIAL: NCT01922167
Title: The Impact of Exercise Training and Leucine Supplementation in Frail Elderly Women With an Exploration Into Mechanistic Explanations
Brief Title: Resistance Exercise Training and Amino Acid Leucine Supplementation in Frail Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jose Morais, Associate Professor and Director, Division of Geriatric Medicine, McGill University; President of the Canadian Geriatrics Society, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MUHC-H-5461
Record Dates: First submitted 2013-07-26; First posted 2013-08-14 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Frail Elderly
Keywords: Aging; Frailty; Leucine; Resistance Exercise
MeSH Terms: conditions — Frailty | interventions — Leucine; Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leucine (Experimental): 2.5 g doses of leucine isolate three times per day (7.5 g total) of leucine, taken by mouth in powder form mixed with liquid for 12 consecutive weeks.
  Interventions: Dietary Supplement: Leucine
- Alanine (Placebo Comparator): 2.5 g doses of alanine isolate three times per day (7.5 g total) of alanine, taken by mouth in powder form mixed with liquid for 12 consecutive weeks.
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Leucine
  Arms: Leucine
Dietary Supplement: Alanine
  Arms: Alanine

SUMMARY:
Frailty is a clinical entity associated with an increase in risk for disease and death and becomes more common as people age. Frailty has a strong relationship with the age-related loss of muscle and strength, termed sarcopenia. Sarcopenia and frailty are strongly associated with disability, especially in women. Adequate protein intake, the amino acid leucine, and resistance exercise training have been individually shown to increase muscle mass to varying degrees. However, no studies have investigated how a longer-term resistance exercise training program with leucine supplementation when protein intake is optimized could increase muscle mass in frail and pre-frail elderly women. In addition, this is the population that stands the most to gain from such an intervention.

The purpose of this study is to investigate the effects of the amino acid leucine added to resistance exercise training on muscle mass and physical performance in frail and pre-frail elderly women with adequate protein intake. We hypothesize that combining leucine in diet with an exercise program would be superior to exercise alone in stimulating muscle protein synthesis and phosphorylation status of muscle cellular key-regulatory proteins, leading to enhanced gains in muscle performance.

A total of 24 subjects will take part in this study, conducted at the McGill University Health Centre (MUHC) Royal Victoria Hospital and the Institut Universitaire de Gériatrie de Montréal (IUGM). All subjects will undergo adjustments to their diet to optimize protein intake and a resistance exercise training program. Half of the participants will receive a supplement of powdered leucine (an amino acid), and the other half of the participants will receive a placebo in the same powder form. Neither the participants nor the study investigators will know which participants are receiving the leucine nor which are receiving the placebo.

Each subjects participation in this study will involve 4 total visits: 2 initial screening visits followed by 2 two-day stays at the Centre for Innovative Medicine (CIM) of the MUHC-Royal Victoria Hospital. These two stays will be spaced by 12 weeks of the intervention (dietary adjustments, resistance exercise training, and the powdered supplement). The two stays each consist of a meal test to assess each subjects metabolic responses to a meal, and to obtain muscle biopsies necessary to measure the rate of protein accumulation in the muscle. Simple physical performance measurements will be taken before and at the completion of the intervention.

This study aims to better understand how the presence of aging affects the body's responses to resistance exercise and how leucine, one of the amino acids that make up proteins, may help build muscle. This in turn, could lead to defining combined diet and exercise strategies to prevent muscle loss often seen with aging.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Examination score > 24
* Time up and go test < 17 s
* Stable weight and diet
* No acute disease
* Body mass index (BMI) 20-35 kg/m^2
* Normal complete blood count (CBC), biochemistry, glycated hemoglobin (A1C), lipid profile, thyroid stimulating hormone (TSH)
* Non-diabetic (Oral Glucose Tolerance Test)
* Negative serology for hepatitis and human immunodeficiency virus (HIV)
* Normal chest X-Ray, electrocardiogram (ECG) and urine analysis
* Non-disabled
* Provide informed consent

Exclusion Criteria:

* Eating disorder,
* Food allergies affecting diet
* Substance abuse
* Active medical conditions including diabetes and any cancer other than skin within 5 years
* Serum creatinine > 110 umol/L, Hb < 110 g/L
* Medications known to interfere with the metabolic endpoint measurements: diuretics, beta-blockers, bronchodilators, non-steroidal anti-inflammatory drugs (NSAIDs), antianginals, antiarrythmics and steroids (other than topical)
* Disability

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-11; Primary Completion 2018-02-08 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Fractional Synthesis Rate (FSR) at 12 weeks | Baseline and at 12 weeks

SECONDARY OUTCOMES:
Change from Baseline in Physical Performance at 12 weeks | Baseline and at 12 weeks
  Short Physical Performance Battery test, Timed-up-and-Go test 6 Minute Walk Test
  1 repetition maximum Hand-grip strength
Change from Baseline in Body Composition at 12 weeks | Baseline and at 12 weeks
  Dual energy X-ray absorptiometry
Change from Baseline in Post-prandial responses at 12 weeks | Baseline and at 12 weeks
  Will measure excursion curves of glucose, insulin, branched chain amino acids, and amino acid profile
Change from Baseline in Fasting levels at 12 weeks | Baseline and at 12 weeks
  Will measure fasting levels of insulin growth factor-1 (IGF-1), interleukin-6 (IL-6), cortisol, as well as resting metabolic rate

OTHER OUTCOMES:
Change from Baseline in Quality of Life at 12 weeks | Baseline and at 12 weeks
  EuroQuol EQ-5D-5L™
Change from Baseline in Mammalian target of rapamycin (mTOR) signalling proteins at 12 weeks | Baseline and at 12 weeks
  Quantity of the following proteins and their phosphorylation status:
  * Protein kinase B (Akt) and phosphorylation on Ser473
  * Eukaryotic translation initiation factor 4E-binding protein 1 (4E-BP1) and phosphorylation on Thr37/46
  * Ribosomal protein S6 kinase beta-1 (S6K1) and phosphorylation on Thr389
  * Ribosomal protein S6 (rpS6) and phosphorylation on Ser240/244
  * Proline-rich Akt substrate of 40 kilodaltons (PRAS40) and phosphorylation on Thr246
  * Forkhead box O3a (FoxO3a) and phosphorylation on Thr32

CONTACTS AND LOCATIONS:
Overall Officials: José A Morais, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Institut Universitaire de Gériatrie de Montréal, Montreal, Quebec
  - Royal Victoria Hospital - Glen Site, Montreal, Quebec

REFERENCES:
- [Derived] Jacob KJ, Sonjak V, Spendiff S, Hepple RT, Chevalier S, Perez A, Morais JA. Mitochondrial Content, but Not Function, Is Altered With a Multimodal Resistance Training Protocol and Adequate Protein Intake in Leucine-Supplemented Pre/Frail Women. Front Nutr. 2021 Jan 22;7:619216. doi: 10.3389/fnut.2020.619216. eCollection 2020. PMID 33553232
- [Derived] Jacob KJ, Chevalier S, Lamarche M, Morais JA. Leucine Supplementation Does Not Alter Insulin Sensitivity in Prefrail and Frail Older Women following a Resistance Training Protocol. J Nutr. 2019 Jun 1;149(6):959-967. doi: 10.1093/jn/nxz038. PMID 31149709